CLINICAL TRIAL: NCT05551078
Title: Thrombophilia Screening in Women After Severe IUGR
Brief Title: Thrombophilia Screening After Severe IUGR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PI102
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: IUGR; Thrombophilia; Pregnancy Complications
MeSH Terms: conditions — Thrombophilia; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women with severe IUGR
  Interventions: Biological: thrombophilia screening

INTERVENTIONS:
Biological: thrombophilia screening — In the IUGR group systematic thrombophilia screening had already been performed.

SUMMARY:
This retrospective study aims to assess the input of thrombophilia screening in pregnant women with severe intra-uterine growth restricted babies.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* Pregnant women
* IUGR defined by an EFW <3rd centile
* IUGR before 25 GW

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: * Women over 18 years old
  * Pregnant women
  * IUGR defined by an EFW <3rd centile
  * IUGR before 25 GW
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Rate of positive's thrombophilia screening | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Matthieu Dap, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided